CLINICAL TRIAL: NCT00264134
Title: A Phase I/II Trial: Docetaxel, Irinotecan, and Carboplatin in the Treatment of Extensive Stage Small Cell Lung Carcinoma
Brief Title: Docetaxel, Irinotecan, and Carboplatin in Extensive Stage Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kentuckiana Cancer Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1047791; CPTAIV-0020-339
Record Dates: First submitted 2005-12-08; First posted 2005-12-12 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Non-small Cell Lung Cancer; Extensive Stage Unresectable
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Irinotecan; Carboplatin

INTERVENTIONS:
Drug: Docetaxel
Drug: Irinotecan
Drug: Carboplatin

SUMMARY:
Primary Objective: To determine the maximum tolerated dose of docetaxel when given with Irinotecan and Carboplatin for the treatment of inoperable lung cancer.

Secondary Objective: To evaluate the dose-related toxicities of this triple regimen in patients with inoperable lung cancer.

DETAILED DESCRIPTION:
A phase I/II dose escalating study to determine the maximum tolerated dose of docetaxel when given with Irinotecan and Carboplatin for the treatment of inoperable lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older unresectable lung cancer measurable or evaluable lesions Karnofsky PS greater than or equal to 60%

Exclusion Criteria:

* untreated CNS metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-06; Study Completion 2005-10

PRIMARY OUTCOMES:
Primary Objective: To determine the maximum tolerated dose of docetaxel when given with Irinotecan and Carboplatin for the treatment of inoperable lung cancer.

SECONDARY OUTCOMES:
Secondary Objective: To evaluate the dose-related toxicities of this triple regimen in patients with inoperable lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Glisson, MD, Principal Investigator — Kentuckiana Cancer Institute
Locations (1):
- Kentuckiana Cancer Institute, Louisville, Kentucky, United States